CLINICAL TRIAL: NCT03387124
Title: Characterization of Stool Consistency and Fecal Microbiota of Breastfed Infants
Brief Title: Breastfeeding Study
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 16.23.INF
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Infant Term Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Breastfed infants — Breastmilk

SUMMARY:
The purpose of this study is to evaluate the stool consistency and microbiota composition of healthy breastfed infants.

DETAILED DESCRIPTION:
This is a prospective, observational, non-interventional study. The purpose of this study is to evaluate the stool consistency and variability in fecal microbiota composition, diversity, and abundance of defined taxa in 75 healthy, term, exclusively breastfed infants. All enrolled infants will participate in the trial for approximately 169 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Infants whose parent(s)/LAR who have reached the legal age of majority in the Philippines
* Infants whose parent(s)/LAR are willing and able to comply with study requirements
* Infants whose parent(s)/LAR who are able to be contacted directly by telephone throughout the study
* Healthy term, singleton infant at birth
* Between 21 to 26 days post-natal age at enrollment visit
* Weight-for-length and head circumference-for-age z-scores are ≥ -3 and ≤ +3 according to WHO Child Growth Standards
* Infants of parent(s)/LAR who have previously made the decision to breastfeed their infant at the time of enrollment

Exclusion Criteria:

* Infants with conditions requiring infant feedings other than those specified in the protocol
* Infants receiving weaning foods or liquids
* Infants who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results
* Infants who are presently receiving or have received medications that could interfere with the interpretation of study results
* Infants or infants whose parent(s)/LAR who cannot be expected to comply with the protocol or with study procedures

Ages: 21 Days to 26 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 75 healthy term exclusively breastfed infants
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Stool Consistency Score | 155 days

SECONDARY OUTCOMES:
Fecal Microbiota Composition | 155 days
Changes in Weight from baseline to 155 days | 155 days
  weight (kg)
Changes in Length from baseline to 155 days | 155 days
  length (cm)
Changes in Head Circumference from baseline to 155 days | 155 days
  head circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira M Estorninos, MD, Principal Investigator — University of Alberta
Locations (1):
- Asian Hospital and Medical Center, City of Muntinlupa, Alabang, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Samuel TM, Hartweg M, Lebumfacil JD, Buluran KB, Lawenko RB, Estorninos EM, Binia A, Sprenger N. Dynamics of human milk oligosaccharides in early lactation and relation with growth and appetitive traits of Filipino breastfed infants. Sci Rep. 2022 Oct 15;12(1):17304. doi: 10.1038/s41598-022-22244-7. PMID 36243744